CLINICAL TRIAL: NCT01340599
Title: Phase II, Randomized, Double Blind, Placebo Controlled Pilot Study of Polyphenon E in Men With Localized Prostate Cancer Scheduled to Undergo Radical Prostatectomy
Brief Title: Defined Green Tea Catechin Extract in Treating Patients With Localized Prostate Cancer Undergoing Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CASE13805; NCI-2011-00606 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-04-20; First posted 2011-04-22 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Stage I Prostate Cancer; Stage IIA Prostate Cancer; Stage IIB Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — polyphenon E; Immunohistochemistry; Immunoenzyme Techniques; Chromatography, High Pressure Liquid; Mass Spectrometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Polyphenon E) (Experimental): Patients receive defined green tea catechin extract PO once daily QD for 4-10 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo radical prostatectomy between days 28-70.
  Interventions: Dietary Supplement: defined green tea catechin extract; Other: immunohistochemistry staining method; Other: immunoenzyme technique; Other: questionnaire administration; Procedure: therapeutic conventional surgery; Other: high performance liquid chromatography; Other: mass spectrometry
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO QD for 4-10 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo radical prostatectomy between days 28-70.
  Interventions: Other: placebo; Other: immunohistochemistry staining method; Other: immunoenzyme technique; Other: questionnaire administration; Procedure: therapeutic conventional surgery; Other: high performance liquid chromatography; Other: mass spectrometry

INTERVENTIONS:
Dietary Supplement: defined green tea catechin extract — Given PO
  Other Names: Polyphenon E
  Arms: Arm I (Polyphenon E)
Other: placebo — Given PO
  Other Names: PLCB
  Arms: Arm II (placebo)
Other: immunohistochemistry staining method — Correlative studies
  Other Names: immunohistochemistry
Other: immunoenzyme technique — Correlative studies
  Other Names: immunoenzyme techniques
Other: questionnaire administration — Ancillary studies
Procedure: therapeutic conventional surgery — Undergo radical prostatectomy
Other: high performance liquid chromatography — Correlative studies
  Other Names: HPLC
Other: mass spectrometry — Correlative studies

SUMMARY:
This randomized pilot phase II trial studies the side effects and how well defined green tea catechin extract works in treating patients with localized prostate cancer undergoing surgery. Defined green tea catechin extract contains ingredients that may prevent or slow the growth of certain cancers.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To evaluate the short-term effects of daily Polyphenon E (defined green tea catechin extract) administration (800 mg epigallocatechin-3-gallate [EGCG] once daily [QD]) during the interval between prostate biopsy and radical prostatectomy (approximately 6 weeks) in men with localized prostate cancer.

II. Compare the change in levels of intermediate biomarkers (Ki-67, B-cell lymphoma 2 [Bcl2], cyclin D, KiP1/P27, vascular endothelial growth factor [VEGF], and cluster of differentiation [CD]31) in biopsy (pre-treatment) and prostatectomy (post-treatment) specimens collected from subjects treated with Polyphenon E or placebo during the period between biopsy and prostatectomy.

III. Compare the change in pre- and post-treatment serum prostate-specific antigen (PSA) level in subjects treated with Polyphenon E or placebo during the period between biopsy and prostatectomy.

IV. Evaluate bioavailability of catechins from Polyphenon E (plasma and tissue catechin levels, catechin metabolites in urine).

V. Evaluate the safety and tolerability of Polyphenon E in this subject population.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive defined green tea catechin extract orally (PO) QD for 4-10 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo radical prostatectomy between days 28-70.

ARM II: Patients receive placebo PO QD for 4-10 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo radical prostatectomy between days 28-70.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Prostate biopsy positive for cancer; clinically localized T1 and T2 stage disease expected, with biopsy specimen available for baseline biomarker measurements
* Scheduled for a radical prostatectomy
* Willing to sign an Institutional Review Board (IRB)-approved informed consent document and adhere to the protocol
* Willing and able to take oral medications
* Willing to refrain from drinking any kind of tea (including herbal tea) or using supplements containing green tea constituents for the duration of the study

Exclusion Criteria:

* Prior hormonal or surgical therapy for prostate cancer; including prior brachytherapy or radiation therapy
* Recent consumption of tea (six or more cups per day) or use of supplements containing green tea within one week of randomization
* Signs or symptoms of progressive or uncontrolled renal, hepatic, hematologic, endocrine, pulmonary, cardiac, neurologic or cerebral disease
* Serum creatinine >= 1.5 x upper limit of normal (ULN)
* Alanine aminotransferase (ALT) >= ULN
* Aspartate aminotransferase (AST) >= ULN
* Alkaline phosphatase (ALP) >= ULN
* Albumin (ALB) =< lower limit of normal (LLN)
* Total bilirubin >= ULN
* Known malignancy at any site within the last five years; with the exception of basal cell carcinoma (BCC)
* Participation in a research trial within the past three months
* Any condition that would interfere with the ability to give informed consent or comply with the study protocol
* Hypersensitivity to tea products or any of the inactive ingredients found in the drug product capsules
* Concomitant use of at least 400 mg per day of a nonsteroidal anti-inflammatory (NSAID) agent two or more times per week

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-10; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Change in levels of intermediate biomarkers in prostate tissue (Ki-67, Bcl2, cyclin D, KiP1/P27, VEGF, and CD31) during treatment with defined green tea catechin extract or placebo during the period between biopsy and prostatectomy | Baseline and at or after 6 weeks of treatment

SECONDARY OUTCOMES:
Changes in the levels of free (f) PSA | After 0, 4, and 6 weeks
  PSA exists in the serum in different molecular forms and that the proportion of "complexed" PSA (PSA-ACT) to "free" PSA(F-PSA) is higher in prostate cancer patients [16]. F-PSA-to-PSA ratio remains constant in men without prostate cancer while total PSA increases. This F-PSA to-PSA ratio is useful diagnostic tool with borderline total PSA values (4.0 to 10.0 ng/mL); additionally values of 20% to 25% F-PSA eliminates 1/3 of biopsies in some studies; and F-PSA of 15.6% and PSA-ACT of 26.7% yielded 95% sensitivity [17]. The F-PSA-to-PSA ratio does not correlate to grade or stage of cancer.
Catechin levels | At baseline, 4 weeks after supplementation, and at time of surgery
  Extraction of Catechins from Prostate Tissue, plasma and urine samples
Number of pts with adverse events as a measure of safety and tolerability | At baseline and every 4 weeks
  AEs will be recorded from the date the informed consent document is signed until the day of surgery. Liver function tests including the Hepatic Function Panel [Alanine Aminotransferase (ALT), Albumin, Alkaline Phosphatase (ALP), Aspartate Aminotransferace (AST), total and direct Bilirubin], as well as amylase and lipase tests will be monitored at baseline and every four (4) weeks for the duration of the study.
Changes in the levels of total (t) PSA | After 0, 4, and 6 weeks
  PSA exists in the serum in different molecular forms and that the proportion of "complexed" PSA (PSA-ACT) to "free" PSA(F-PSA) is higher in prostate cancer patients [16]. F-PSA-to-PSA ratio remains constant in men without prostate cancer while total PSA increases. This F-PSA to-PSA ratio is useful diagnostic tool with borderline total PSA values (4.0 to 10.0 ng/mL); additionally values of 20% to 25% F-PSA eliminates 1/3 of biopsies in some studies; and F-PSA of 15.6% and PSA-ACT of 26.7% yielded 95% sensitivity [17]. The F-PSA-to-PSA ratio does not correlate to grade or stage of cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Gupta, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States